CLINICAL TRIAL: NCT06649708
Title: A Phase I/IIa, First-in-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of HX044 in Patients with Advanced Solid Tumor Malignancies
Brief Title: HX044,FIH Study in Patients with Advanced Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanx Biopharmaceuticals (Wuhan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Hangzhou Hanx Biopharmaceuticals, Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX044-I-01
Record Dates: First submitted 2024-10-03; First posted 2024-10-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HX044 (Experimental): Conventional dose-escalation design with 3+3 cohort size. Patients received HX044 treatment at assigned dose level on a Q3 weekly basis.
  Interventions: Drug: HX044

INTERVENTIONS:
Drug: HX044 — Conventional dose-escalation design with 3+3 cohort size. All administered on a Q3 weekly basis. Dose escalation will be based on the absence of DLTs during the 21-day DLT evaluation after a review of safety data by the Safety Review Escalation Committee. Subjects will continue on study treatment until the subject develops an intolerable toxicity, withdraws consent, develops progression of disease, death, lost to follow-up, start of new anticancer treatment or up to study treatment duration of 24 months, whichever comes first.

SUMMARY:
The study will consist of a dose-escalation and dose-expansion component to establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D), and to evaluate the preliminary antitumor activity of HX044.

HX044 is an investigational drug that has not yet been approved by the Food and Drug Administration (FDA) or any other regulatory authorities for commercial purposes. This is the first study in which HX044 will be given to humans. The study drug has been tested in animals and was found to be well-tolerated with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate by providing written informed consent and agreeing to comply with protocol and scheduled visit;
2. Male or female subject aged 18-75 years, inclusive;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
4. Histologically confirmed advanced malignant solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.
5. At least 1 measurable tumor (It is acceptable to allow patients with no measurable lesion but evaluable tumor lesion in the first 2 dose levels in Phase I and at least 1 measurable tumor lesion must be present in Phase IIa) according to RECIST v1.1
6. Life expectancy ≥ 12 weeks.
7. Adequate organ function, as indicated by the following laboratory values: •Hematology (no growth factor and blood transfusion are allowed within 14 days before start of first dose study treatment): Hemoglobin ≥90g/L Absolute neutrophil count ≥1.5×109/L Platelet count ≥100×109/L

   * Hepatic: Serum total bilirubin ≤1.5 × upper limit of normal (ULN); or direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 × ULN
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (ALT and AST ≤ 5 × ULN for subjects with liver metastases)
   * Renal:Serum creatinine ≤1.5 × ULN
   * Coagulation: Prothrombin time/international normalized ratio ≤1.5 × ULN or activated partial thromboplastin time ≤ 1.5 × ULN (for subjects on anticoagulants, prothrombin time or activated partial thromboplastin time must be within the normal range foranticoagulants).

Exclusion Criteria:

1. Prior malignancy active within the previous 5 years except for the tumor for which a subject is enrolled in the study and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
2. Receipt of any anticancer (chemotherapy, radiation therapy, investigational drugs including small molecular inhibitors, endocrine therapy, immunotherapy) therapy within 4 weeks prior to the first dose of study treatment or 5 half-lives of the therapy, whichever is shorter.
3. Severe cardiovascular disease including symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina, uncontrolled hypertension, cardiac arrhythmia, a history of myocardial infarction within 6 months or a history of arterial thromboembolic event and pulmonary embolism within 3 months of the first dose of investigational agent, as follows:

   * QT/QTc interval prolongation (using Fredericia's QT correction formula) at baseline, Female > 470 ms, Male > 450 ms;
   * Medications to prolong the QT/QTc interval are currently being taken;
   * Family history of long QT syndrome.
4. Patients with a history of or presently experiencing an active autoimmune disease within 2 years of initiating study drug, or those who are at high risk of relapse ; however, subjects with the following are allowed to enroll:

   * Type I diabetes that is stable after a fixed dose of insulin or other hypoglycemic;
   * Only requiring hormone replacement therapy for autoimmune hypothyroidism;
   * Skin disease that does not require systemic treatment such as eczema rash that accounts for <10% of the body surface, psoriasis without ophthalmic symptoms.
5. Subjects who received any major surgery within 4 weeks before the first dose of study treatment (except for diagnostic surgery), and/or subjects who may require major surgery during the study.
6. Lung diseases such as, interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, interstitial pneumonia. Patients with well controlled chronic obstructive pulmonary disease (COPD) are allowed.
7. Subjects with primary central nervous system (CNS) malignancies, symptomatic CNS metastases, symptomatic parenchymal brain leptomeningeal disease or spinal cord compression, except for the following: who has received prior treatment (surgery/radiotherapy) before signing informed consent form (ICF) and is clinically stable for at least 3 months is allowed (prior treatment with corticosteroids are permitted but must stop 14 days before commencing study treatment）
8. Use of any live vaccines within 4 weeks before the first dose of study treatment.
9. A history of psychotropic substance abuse who is unable to quit.
10. Any patient with an uncontrolled illness such as cardiovascular and cerebrovascular diseases, diabetes, high blood pressure, et, and other severe, acute or chronic medical or psychiatric diseases or laboratory abnormalities that, in the Investigator's opinion, may increase the study-related risks or interfere with the interpretation of the findings.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) | All AEs up to 90(±7）days after the last dose of study treatment
  An AE is any untoward medical occurence in a patient or subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of Participants With Dose-Limiting Toxicities(DLT) of HX044 | At the end of Cycle 2(each cycle is 21±3 days)
  All AEs/toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events,Vesion5.0(NCI CTCAE v5.0);For the purpose of dose escalation, any of the following AEs occurring during the DLT observation period that were attributable to one or both study drugs were classified as DLTs.

SECONDARY OUTCOMES:
Objective response rate (ORR) per Investigator Assessment Using RECIST 1.1 and iRECIST | Approximately 2 years
  Objective response rate (ORR) ,using RECIST 1.1 and iRECIST criteria, is defined as the proportion of subjects with best overall response of complete response(CR)/iCR or partial response(PR)/iPR after treatment.
Disease control rate(DCR) per Investigator Assessment Using RECIST 1.1 and iRECIST | Approximately 2 years
  Disease control rate(DCR) ,using RECIST 1.1 and iRECIST criteria, is defined as the proportion of subjects with best overall response of complete response(CR)/iCR or partial response(PR)/iPR or disease stabilization(SD)/iSD after treatment.
Number of participants with positive Anti-Drug Antibody(ADA) of HX044 | Cycle 1,2,3,4,5,6,10,14,18 and then every 8 cycles,Day 1: with 60 minutes before the start of the infusion.
  ADA blood samples are assayed for anti-HX044 antibodies.
Time of Cmax(Tamx) of HX044 | Approximately 2 years
  Time to reach HX044 maximum observed serum concentration
Terminal Half life( t½) of HX044 | Approximately 2 years
  HX044 terminal half-life.
Area Under the serum concentration-time curve(AUC) | Approximately 2 years
  HX044 area under the serum concentration-time curve

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Blacktown Hospital, Blacktown, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Cabrini Health Limited, Malvern, Victoria

IPD SHARING:
Plan to Share IPD: No